CLINICAL TRIAL: NCT04363606
Title: Chronic Fatigue Etiology and Recovery in Covid-19 Patients : the Role of Fatigability and Stay in Intensive Care
Brief Title: Chronic Fatigue Etiology and Recovery in Covid-19 Patients: the Role of Fatigability
Acronym: FatCovid-19
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: under-inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: University of Saint-Etienne (Unknown); Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20CH085; 2020-A00982-37 (Other: ANSM)
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Chronic Fatigue Syndrome; Intensive Care Unit; Muscle
Keywords: Neuromuscular function; Fatigability
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Surveys and Questionnaires; Hematologic Tests; Actigraphy; Occult Blood; Diet Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- "Non-fatigued" patients who have been in intensive care units (Experimental)
  Interventions: Other: Questionnaires; Biological: blood test; Other: Maximal effort test; Device: actigraphy; Device: Neuromuscular evaluation; Other: stool analysis; Other: food diary
- "Fatigued" patients who have been in intensive care units (Experimental)
  Interventions: Other: Questionnaires; Biological: blood test; Other: Maximal effort test; Device: actigraphy; Device: Neuromuscular evaluation; Other: stool analysis; Other: food diary
- patients who have not been in intensive care units (Experimental)
  Interventions: Other: Questionnaires; Biological: blood test; Other: Maximal effort test; Device: actigraphy; Device: Neuromuscular evaluation; Other: stool analysis; Other: food diary

INTERVENTIONS:
Other: Questionnaires — Quality of life Depression Physical pain Social provisions Quality of sleep
Biological: blood test — complete blood count and cytokine concentration, TNF-alpha, LDL oxidized, AOPP, SOD, GPX, catalase, albumin, transthyretin, RBP, transferin, α-1 glycoprotein acide, ferritine, selenium, zinc, magnesium
Other: Maximal effort test — The maximal effort test with VO2max recordings will be assessed during the first visit to the laboratory.
Device: actigraphy — assessment of sleep quality
Device: Neuromuscular evaluation — * The maximum isometric force produced by the knee extensors will be measured on the ergometer
  * the intensity of muscular electrical activity recorded by surface electromyography
  * Peripheral nerve stimulation
  * Transcranial magnetic stimulation
  * Magnetic resonance imaging
Other: stool analysis — analyze the composition of the intestinal microbiote. concerns only the patients of Saint Etienne
Other: food diary — 3 days of information to determine nutrient intakes. concerns only the patients of Saint Etienne

SUMMARY:
Chronic fatigue is the most common and debilitating symptom in intensive care unit (ICU) survivors. Indeed, it has been widely reported that patients who stayed in ICU for prolonged periods report a feeling of tiredness for months to years after ICU discharge. This symptom seems particularly pronounced in Covid-19 patients and may affect their quality of life by decreasing their capacity to perform simple tasks of daily life.

The aim of the present project is to determine whether deteriorated neuromuscular function (i.e. increased fatigability) is involved in the feeling of fatigue of Covid-19 patients. Because the causes of this feeling are multi-dimensional, a large battery of tests will allow us to better understand the origin of chronic fatigue. A better knowledge of chronic fatigue etiology and its recovery will allow to optimize rehabilitation treatments to shorten the persistence of chronic fatigue and in fine improve life quality.

ELIGIBILITY:
Inclusion Criteria for patients who have been in intensive care :

* Diagnosed with Covid-19
* Ventilated in ICU for at least 3 consecutive days
* ICU discharge between 4 and 8 weeks
* Approval received from a physician
* Command of the French language

Inclusion Criteria for patients who have NOT been in intensive care :

* Diagnosed with Covid-19 : positive serological test or positive PCR test following nasopharyngeal swabbing
* Approval received from a physician
* Command of the French language

Exclusion Criteria:

* Taking neuroactive substances that can alter corticospinal excitability
* Patients with co-morbidities leading to significant fatigue: e.g. cancerous pathologies, sleep apnea
* Patients with neurodegenerative or neuromuscular disease
* Contraindication to the application of a magnetic field
* Contraindication to the practice of Magnetic Resonance Imaging
* Participant is pregnant
* Patients with psychiatric disorders
* Paraplegic and hemiplegic patients
* Addictive disorders

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
voluntary maximum force reduction | 6 weeks post-discharge

SECONDARY OUTCOMES:
Neuromuscular function : cortical activity | 6 weeks post-discharge
  Level of cortical activation and cortico-spinal excitability measured by transcranial magnetic stimulation
Neuromuscular function : Peripheral function | 6 weeks post-discharge
  Peripheral function by electrical nerve stimulation
Maximal oxygen uptake (VO2max) | 6 weeks post-discharge
  measured by effort test
quality of sleep | 6 weeks post-discharge
  measured by actigraphy
muscle volume | 6 weeks post-discharge
  with Magnetic resonance imaging
metabolic fatigue | 6 weeks post-discharge
  measured by a Phosphorus 31 Nuclear magnetic resonance test
microbiote intestinal | baseline and 6 months
  stool analysis (concerns only the patients of Saint Etienne)

CONTACTS AND LOCATIONS:
Overall Officials: Jérome MOREL, MD PhD, Principal Investigator — CHU de Saint Etienne
Locations (8):
- France (8):
  - CHU de Grenoble, Grenoble
  - Clinique de la Sauvegarde - Lyon, Lyon
  - Hôpital Croix Rousse - HCL, Lyon
  - Centre Hospitalier de Lyon Sud, Pierre-Bénite
  - Hôpital privé de la Loire, Saint-Etienne
  - Chu Saint-Etienne, Saint-Etienne
  - Clinique Mutualiste Saint Etienne, Saint-Etienne
  - Hôpital Henry Gabrielle, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kennouche D, Foschia C, Brownstein CG, Lapole T, Rimaud D, Royer N, LE Mat F, Thiery G, Gauthier V, Giraux P, Oujamaa L, Sorg M, Verges S, Doutreleau S, Marillier M, Prudent M, Bitker L, Feasson L, Gergele L, Stauffer E, Guichon C, Gondin J, Morel J, Millet GY. Factors Associated with Fatigue in COVID-19 ICU Survivors. Med Sci Sports Exerc. 2024 Sep 1;56(9):1563-1573. doi: 10.1249/MSS.0000000000003455. Epub 2024 Apr 14. PMID 38742855